CLINICAL TRIAL: NCT03975179
Title: A Randomized Controlled Trial for Doing vs. Omitting Intraoperative Frozen Section Biopsy For Resection MArgin Status in Selected Patients Undergoing Breast Conserving Surgery
Brief Title: Omitting vs. Doing Intraoperative Frozen Section Biopsy for Margin Status in Breast Conserving Surgery
Acronym: OFF-MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Breast Cancer Study Group (Other)
Responsible Party: Principal Investigator, Byung Joo Chae, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC19EEDT0031
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: frozen section biopsy; resection margin; breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frozen section omission (Experimental): Intraoperative frozen section biopsy of resection margin will not be performed
  Interventions: Procedure: Omission of intraoperative frozen section biopsy for margin status
- Frozen section (Active Comparator): Intraoperative frozen section biopsy of resection margin will be performed. Margin evaluation of superior, medial, lateral, inferior margin is recommended but will follow surgeon's discretion.
  Interventions: Procedure: Frozen section biopsy for margin status

INTERVENTIONS:
Procedure: Omission of intraoperative frozen section biopsy for margin status — Omitting intraoperative frozen section biopsy for margin status in patients undergoing breast conserving surgery
  Arms: Frozen section omission
Procedure: Frozen section biopsy for margin status — Performing intraoperative frozen section biopsy for margin status in patients undergoing breast conserving surgery
  Arms: Frozen section

SUMMARY:
* Study phase: 3
* Indication: Breast cancer patients undergoing breast conserving surgery
* Primary objectives: To determine the effect of selective omission of intraoperative margin evaluation via frozen section on margin positive rate Secondary objectives: To determine the effect of selective omission of intraoperative margin evaluation via frozen section on reoperation rate, local recurrence rate, operation time, resection volume, medical cost and patient quality-of life
* Hypothesis: Omitting intraoperative margin evaluation via frozen section biopsy in selected breast cancer patients does not increase margin positive rate
* Study design: Randomized controlled trial
* Sample size: 1292 patients
* Procedures: breast conserving surgery +/- margin frozen section biopsy (+/- additional resection)

DETAILED DESCRIPTION:
1.1 Preoperative work-up Preoperative breast MRI is recommended to assess multifocal/centric lesions and non-mass enhancement surrounding main mass. Preoperative needle localization or skin marking is done by each hospital's method.

1.2 Surgical procedure Initial wide excision is performed as usual. The recommended target gross margin is one finger breadth. Orientation of the specimen will be done according to each center's principle. Randomization for frozen section biopsy vs. omission is done intraoperatively, after initial wide excision. For the frozen section biopsy omission group, no further procedures will be done. For the frozen section biopsy group, frozen section biopsy is performed on the specimen or cavity by the operating surgeon. The precise method is decided by the surgeon's discretion, but the recommended method is as follows. A minimum 1 x 0.5cm size of breast parenchymal tissue will be excised at minimum four directions of the specimen or cavity with a thickness of approximately 0.1cm (Figure).

Additional resection according to frozen section biopsy result will be decided by the surgeon's discretion. After review of final pathology report, decision of second operation for re-excision will also be done by surgeon's discretion. A recommendation of considering re-excision for only a positive margin (tumor on inked margin) is noted but not mandatory. Data on additional resection or re-excision must all be reported.

1.3 Pathology procedure Evaluation procedure of the frozen section biopsy specimen and wide excision, additional excision specimen is done by each hospital's method. A pathology report of both intraoperative frozen section biopsy result and final pathology result of the frozen section biopsy tissue must be done. Gross specimen measurements (height x length x depth) must be specified on pathology report. Also margin status must be recorded, positive margin defined as "no ink on tumor" for DCIS and invasive cancer. Recording of margin distance from superior, inferior, medial, lateral, margin is recommended. If all margin distance is not feasible for recording, at least margin distance of closest margin must be recorded. The final pathology result of the additional resection specimen after frozen section result must describe whether residual cancer cells were present and the site of them. This is the same for re-operation resection specimens. Thorough microscopic examination for residual cancer cells in additional/re-operation resection specimens is warranted.

1.4 Postoperative care and adjuvant therapy Postoperative care will be performed as usual. Routine adjuvant care will be given, including adjuvant radiation therapy.

1.5 Follow-up The subject's participation of this clinical trial finishes at last fill in of postoperative quality-of-life questionnaire or after last surgery.

Annual clinical examination, mammography and breast sonography is recommended for 5-year local recurrence assessment. Local recurrence is defined as pathologically confirmed ipsilateral breast tumor recurrence.

1.6 Alternatives This is a randomization between two commonly accepted surgical techniques and there is not any oncological increased risk with either. All routine precautions will be taken to minimize overall surgical risk. Alternatives to the trial would be to have standard breast conserving surgery with or without intraoperative frozen section biopsy according to surgeon's discretion and patients will be informed of this. In addition, all patients will be informed of their option for mastectomy as well.

1.7 Compensation Patients will not be paid for participating in this study. Medical expenses occurred during this study will be paid by the patient. This includes costs associated with re-operation for margin re-excision.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer by core needle biopsy with clinical stage T1-3 by American Joint Committee on Cancer(AJCC) 8th edition
* Candidate of breast-conserving surgery
* Daughter nodule within ≤ 1cm distance of main mass on breast MRI
* Non-mass enhancement extent within ≤ 1cm distance of main mass on breast MRI
* Ability to understand and willing to sign a written informed consent document : Patients who consent about deciding whether frozen biopsy will be performed by randomization

Exclusion Criteria:

* cT4 tumors (AJCC 8th edition)
* Cancer diagnosis confirmed by vacuum-assisted biopsy or surgical biopsy
* Initial operation plan being total mastectomy (conversion to total mastectomy after intraoperative frozen section biopsy is acceptable)
* Personal history of ipsilateral breast cancer
* Ductal carcinoma in situ component on CNB result
* Lobular carcinoma (invasive, in situ)
* Neoadjuvant chemotherapy
* Lesion with microcalcification (microcalcification that is only contained inside the cancer mass is acceptable)
* Multicentric tumor, however a daughter nodule within ≤ 1cm distance on breast MRI is acceptable
* Non-mass enhancement extent wider than 1cm distance of main mass on breast MRI

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1292 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Resection margin status | 2 weeks after primary surgery
  Margin status data will be obtained from pathology report. Positive margin is defined as "no ink on tumor" for DCIS and invasive cancer. A close margin of any distance is defined as a negative margin

SECONDARY OUTCOMES:
Reoperation rate | 2 months after primary surgery
  Additional operation for re-excision of margin is defined as a reoperation. The decision for a reoperation is determined by the surgeon. Data regarding reoperation and reason for reoperation must be recorded.
Operation time | Immediately after primary surgery
  Operation time is defined by time from incision to closure, which will be obtained from anesthesia report.
Cost effectiveness | 3 months after primary surgery
  Data for in-hospital cost including cost for re-excision will be collected. Opportunity cost due to elongated surgery time and labor costs from the pathology department will also be calculated and included.
Resection volume | 3 months after primary surgery
  Resected volume is calculated from gross specimen measurements of pathology report (volume = width/2 * height/2 * depth/2). When additional resection is performed, resected volumes are reported separately.
Number of patients with residual cancer after reoperation | 3 months after primary surgery
  Whether residual cancer cells are present in re-operation specimens for excision of resection margin. Thorough microscopic examinations are warranted for this endpoint.
Number of patients with residual cancer after re-excision according to frozen section biopsy result | 3 months after primary surgery
  Whether residual cancer cells are present in additional resection specimens performed according to frozen section biopsy result of resection margin. Thorough microscopic examinations are warranted for this endpoint.
Patient quality-of-life assessment: BREAST-Q survey | 1 year after primary surgery
  Quality-of-life assessment is performed by using the Korean version of the BREAST-Q survey for breast conserving therapy which is a questionnaire for patient reported outcome measurement. An assessment for physical well-being, psychosocial well-being, sexual well-being, satisfaction with breasts/outcome/care will be done. Each subscale will be reported with a scale of 0 - 100. A higher value is considered a better outcome. No total score will be calculated.
  The survey module is filled out pre- and post-operatively. Postoperative module is scored 1 month postoperatively (within one month of date of final operation but before start of radiotherapy) and within 2 months of completion of radiotherapy.

OTHER OUTCOMES:
Local recurrence | 5 years after primary surgery
  Local recurrence is defined as pathologically defined ipsilateral breast tumor recurrence. Median follow up period is 5 years. Annual clinical examination, mammography and breast sonography is warranted for evaluation of local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Byung Joo Chae, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Ilsan Paik Hospital, Goyang-si
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Raw data can be shared among co-investigators after deidentification of personal information of participated patients under request to PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of recruitment - 10 years after end of trial
Access Criteria: co-investigators

REFERENCES:
- [Derived] Yoo TK, Kang YJ, Jeong J, Song JY, Kang SH, Lee HY, Kim ET, Yi O, Lee HB, Choi S, Park HS, Gwak G, Kim JI, Kim MK, Lee J, Kang HJ, Chae BJ. A Randomized Controlled Trial for Doing vs. Omitting Intraoperative Frozen Section Biopsy for Resection Margin Status in Selected Patients Undergoing Breast-Conserving Surgery (OFF-MAP Trial). J Breast Cancer. 2021 Dec;24(6):569-577. doi: 10.4048/jbc.2021.24.e51. PMID 34979601